CLINICAL TRIAL: NCT07361601
Title: Implementation of Aging in Place Services for Older Adults With Alzheimer's Disease
Brief Title: Implementation of AIP Services for Older Adults With AD
Acronym: PYL-AIP
Status: Not yet recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Lee Lindquist, Professor of Medicine, Section Chief - Geriatrics, Northwestern University
Other Study IDs: R01AG091323-01
Record Dates: First submitted 2026-01-21; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
Keywords: Aging in place; Long term care planning
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will longitudinally follow a cohort of older adults to better understand how decisions about aging in place or transitioning to long-term care-and the implementation of those decisions-are influenced by age-related changes (e.g., cognition, health literacy, chronic conditions) and social supports (e.g., caregivers).

DETAILED DESCRIPTION:
Participants currently enrolled in the National Institute on Aging (NIA)-funded study Decision Making and Implementation of Aging-in-Place/Long-Term Care Plans Among Older Adults (R01AG058777) will continue to be followed for an additional 42 months.

This study will examine how decision-making and planning related to aging in place change over time and how these processes are influenced by age-related changes (e.g., cognition, multiple chronic conditions), social influences (e.g., adult children, spouses, friends), and environmental factors (e.g., rural vs. urban residence, housing type). The study will also assess whether aging-in-place planning translates into timely implementation of services and whether implemented plans are concordant with the goals and preferences of older adults and their surrogate or caregiver decision makers.

In addition, the study will examine how age-related changes, social influences, and environmental factors interact to affect planning and implementation of aging-in-place and long-term care decisions over time.

ELIGIBILITY:
Inclusion Criteria - Current Cohort:

1. Active participant in the 'Decision Making and Implementation of Aging-in-Place/Long Term Care Plans among Older Adults' [R01AG058777] study;
2. Age 65 years or older (older adult); age 18 years or older (caregiver)
3. Speak English; and
4. Pass UBACC (University of California, San Diego Brief Assessment of Capacity to Consent) cognitive assessment

Inclusion Criteria - Caregiver:

1. Age 18 years or older;
2. Speak English;
3. Currently assist enrolled, older adult study participant with activities such as managing their health, and/or household activities (i.e., taking them to the doctor, housekeeping, meal prep, medication reminders); and
4. Pass UBACC (University of California, San Diego Brief Assessment of Capacity to Consent) cognitive assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of a cohort of older adults who are currently enrolled in the longitudinal study, R01AG058777. Older adults as well as their caregivers, where appropriate, are being followed over time to assess decision-making and planning related to aging in place and potential transitions to long-term care. The cohort includes individuals with varying levels of cognitive function, health status, chronic conditions, and social support, as well as diverse living environments (e.g., rural and urban settings, different types of housing). Participants will continue to be followed prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 285 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of participant long term care planning for Alzheimer's Dementia/Memory Loss | Assessed every 6 months, 108 months reported
  Participants are asked "If you developed Alzheimer's or memory loss and could no longer live independently in your home, have you decided what your living preferences (e.g. stay in own home, retirement/long term care community) would be?" Decision-making is measured as a binary ('yes', 'no') outcome at each time-point. Will report % of participants who indicated "YES", that they have decided on their living preferences. Frequencies given for 108 month timepoint per primary outcome analysis.

SECONDARY OUTCOMES:
Rate of participant planning for in-home care in the event of Alzheimer's Disease/Memory Loss | Assessed every 6 months, 108 months reported
  Participants are asked "Have you already decided what your preferences would be if you developed Alzheimer's Disease or memory loss and needed caregiver help in your home?". Responses recorded as binary. Will report % of participants who indicated "YES", that they have decided on their caregiver preferences. Frequencies given for 108 month timepoint per primary outcome analysis.
Rate of participant planning for memory care in the event of Alzheimer's Disease/Memory Loss | Assessed every 6 months, 108 months reported
  Participants are asked "Have you decided what your long-term care preferences (e.g. where you would prefer to go if you needed to be in a nursing home or memory care), would be if you ever developed Alzheimer's Disease or memory loss? " Here, participants were specifically asked about "memory care" vs other types of care options. Responses recorded as binary. Will report % of participants who indicated "YES", that they have a plan for that scenario. All statistical analyses for this outcome will reflect data at the 108 month assessment.
Rate of participant planning for a hospitalization requiring rehabilitation outside the home | Assessed every 6 months, 108 months reported
  Participants are asked "Have you already decided what your preferences would be if you were hospitalized and needed post-hospitalization rehabilitation outside of the home? " Responses recorded as binary. Will report % of participants who reported positively ("Yes") that they had a plan for the scenario. Frequencies given for 108 month timepoint per primary outcome analysis.
Rate of participant planning for a hospitalization requiring in-home care | Assessed every 6 months, 108 months reported
  Participants are asked "Have you already decided what your preferences would be if you were hospitalized and needed caregiver help in your home?" Responses recorded as binary. Will report % of participants who reported positively ("Yes") that they had a plan for the scenario. All statistical analyses for this outcome will reflect data at the 108 month assessment.
Rate of participant decision-making contemplation: Alzheimer's Dementia/Memory Loss (ADML) | Assessed every 6 months, 108 months reported
  Participants are asked a panel of statements about contemplation for decision-making in the event of Alzheimer's Dementia/Memory Loss (ADML). Participants are shown a statement and asked to gauge how frequently they contemplated the possibility of the given scenario, ranging from "Never" to "A Lot". Frequencies given for 108 month timepoint per primary outcome analysis. Each statement is prefixed by "How much have you thought about..."
Rate of participant decision-making contemplation: Hospitalization | Assessed every 6 months, 108 months reported
  Participants were asked a panel of statements about contemplation for decision-making in the event of Hospitalization. Participants are shown a statement and asked to gauge how frequently they contemplated the possibility of the given scenario, ranging from "Never" to "A lot". Frequencies given for 108 month timepoint per primary outcome analysis. Each statement is prefixed by "How much have you thought about..."
Participant utilization of long-term care services (RUI) | 72-month timepoint
  Participant utilization of long-term care services such as in-home caregivers as measured by the Resource Use Inventory (RUI). Frequencies provided for "yes" responses to individual items on the inventory. This outcome measure collected as part of the LitCog assessment battery. Frequencies reflect all available data at the 72 month assessment.
Previous health experiences: Self and others | 72-month timepoint
  Participants are asked a panel of non-validated questions about their previous health experiences and their experiences with others. Frequencies reflect all available data at the 72 month assessment.
Event and Goal Concordance | Assessed every 6 months, 108 months reported
  Participants report on any hospitalizations, recent memory loss, and changes in lifestyle due to hospitalization and memory loss. Responses are binary (yes/no), with a N/A and "unsure/don't know" option. Questions are non-validated. Frequencies given for 108 month timepoint per primary outcome analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Lee A Lindquist, MD MPH MBA, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD and related data dictionaries available.